CLINICAL TRIAL: NCT04654273
Title: EX-PO Trial : Evaluation of the Occlusion Pressure (PO.1) in Extubation Failure
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: EX-PO
Record Dates: First submitted 2020-11-29; First posted 2020-12-04 (Actual); Last update posted 2021-07-08 (Actual); Status verified 2021-01

CONDITIONS: Respiratory Failure
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Measuring bedside occlusion pressure in neurosurgical or surgical critically ill patients could tell us about the patient's respiratory drive, and therefore, tell us whether or not extubation will be successful.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old,
* Hospitalized in surgical or neurosurgical intensive care units
* Patients under mechanical ventilation for more than 48 hours,
* Meeting the criteria for severability (spontaneous ventilation test),
* Free subject, without tutorship or curatorship or subordination,
* Patients benefiting from a Social Security scheme or benefiting through the intermediary of a third party,
* No objection given by the patient and / or relative after clear and fair information about the study.

Exclusion Criteria:

* Tracheostomized patients,
* Persons benefiting from enhanced protection, namely minors, persons deprived of their liberty by a judicial or administrative decision, persons staying in a health or social establishment, adults under legal protection,
* Pregnant and / or lactating women.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients hospitalized in surgical or neurosurgical intensive care units of CHU de Poitiers, under mechanical ventilation for more than 48 hours, meeting the criteria for severability.
Sampling Method: Probability Sample
Enrollment: 152 (Estimated)
Dates: Start 2020-11-30 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-01-31 (Estimated)

PRIMARY OUTCOMES:
Number of re-intubations after extubation | 7 days

CONTACTS AND LOCATIONS:
Locations (1):
- CHU POitiers, Poitiers, France